CLINICAL TRIAL: NCT06743971
Title: 0-3 Months Infantile Colic The Effect of Ocean Sound on Babies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, ÖZLEM YÜKSEL ALTUNTAŞ, Nurse, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OALTUNTAS
Record Dates: First submitted 2024-06-10; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Infantile Colic
Keywords: pediatric nurse; infantil colic; cry; sleep
MeSH Terms: conditions — Colic; Crying

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Parents will let their babies listen to ocean sounds during colic cries for 1 week.
  Interventions: Behavioral: ocean sound concert
- control (No Intervention): Parents will continue with routine care practices during the baby's colicky cries

INTERVENTIONS:
Behavioral: ocean sound concert — intervention group listened to the ocean sound, the control group continued their daily care routines
  Arms: experimental

SUMMARY:
Infant colic is one of the most common health problems in newborns and infants. It is a syndrome of unknown cause, occurring in attacks, weakened by clenched fists, hardening of the abdomen, flatulence, pulling the legs to the abdomen, very difficult to stop and excessive crying. Various studies have been conducted on this subject and the incidence rates in healthy babies vary between 10-40%. Significant behavioral problems may arise in sleep, rest and feeding due to frequent and prolonged periods of arrest, which are considered to be the upper point of normal crying. In these mothers, symptoms such as helplessness, fatigue, insomnia, exhaustion, loss of life, feelings of inadequacy, anxiety and crying problems may occur. In these mothers, variability is also extended. While in the womb, the fetus is attuned to the sound of the blood in the mother's arteries and the rocking motion of her abdomen. During infancy, the uterus is constantly hearing sounds at a higher frequency than a vacuum cleaner and these sounds stimulate a calming reflex in the baby. Our aim in this study was to investigate the sound of the ocean in infants with infantile colic aged 0-3 months.

DETAILED DESCRIPTION:
Infantile colic is one of the most common health problems in the neonatal and infancy periods. It is a syndrome of unknown cause, occurring in attacks, characterized by clenched fists, abdominal hardening, flatulence, pulling the legs to the abdomen, and excessive crying that is very difficult to stop.

Although there are different definitions of colic, according to Wessel's rule of thirds definition, which is the most widely accepted and accepted as a diagnostic criterion in most studies, unexplained and uncontrollable crying spells with onset in the first weeks, usually in the first 3 months, lasting more than 3 hours a day, more than 3 days a week and at least 3 weeks, usually occurring in the afternoon and evening hours are accepted as gas pains .

Various studies have been conducted on this subject and the incidence in healthy infants has been found to be between 10-40%.

Studies have reported that colic symptoms disappeared at the end of the 4th month in 90% of cases. Important behavioral problems may arise in the baby's sleep, rest and feeding due to frequent and prolonged crying bouts of the baby, which are considered the upper point of normal crying.

This may lead to symptoms such as helplessness, fatigue, insomnia, exhaustion, loss of self-confidence, feelings of inadequacy, anxiety and breastfeeding problems. Studies have shown that the frequency of depression also increases in these mothers.

The frequency of colic does not show any difference between boys and girls, breastfed or formula-fed infants, term and preterm infants. It has been reported that colic is associated with marital problems, parental stress perception, lack of parental self-confidence during pregnancy, dissatisfaction with childbirth and family stress levels. Colic is a condition that needs to be managed well because it causes stress in the mother and physician as well as the baby, causes anxiety and depression in the mother, causes breastfeeding to be interrupted and formula to be given instead of breast milk, and increased risk of battering.

Although the causes of colic cannot be fully explained, factors such as food allergy or lactose intolerance, hypersensitivity, abnormal peristalsis or excessive gas, tension and stress in the family, bottle feeding or swallowing air during excessive crying, gastro-esophageal reflux, low birth weight, psychosocial problems in the mother are thought to cause colic. Since the cause is not known exactly, there is no definitive treatment. Some treatment methods are recommended to relieve symptoms. These symptomatic treatment methods include medication, diet and behavioral approaches.

Transition from the womb to the outside world is a very challenging situation for the child. Leaving the mother's womb, where all needs are met, and coming into the world, needing someone else to survive, can be a complete shock for the baby. While some babies adapt easily, others cannot.

Hearing is the baby's ability to distinguish sounds of different frequency, intensity and duration. It is an important sensory experience that begins in the intrauterine period and can lead to physiological and behavioral consequences throughout life.

This may lead to symptoms such as helplessness, fatigue, insomnia, exhaustion, loss of self-confidence, feelings of inadequacy, anxiety and breastfeeding problems. Studies have also shown that the frequency of depression increases in these mothers. One of these scientists, Dr. Harvey Karp, is the scientist who says that there are some things that can be done to make the baby feel as if he/she is in the womb after coming home.

While in the womb, the fetus is habituated to the sound of blood in the mother's arteries and the rocking motion of the abdomen. While in the uterus, the fetus constantly hears sounds with a frequency higher than that of a vacuum cleaner, which stimulate a calming reflex in the fetus.

Music is a natural method used in pain management because of its ease of use. The mechanism by which music therapy relieves pain is not known exactly. It is thought to have a relaxation or distraction effect. Many babies can be calmed by the sound of a fan or vacuum cleaner, tape recordings of the rumblings heard in the womb, sounds in nature or their fathers' voices.

In experiments, it was observed that newborn babies lying in a room where the sound of the uterus was played on a tape recorder fell asleep earlier than babies lying in a room where no sound was played. This is considered to be an indication that newborns begin to gain a certain sensitivity to music before they are born.

The aim of this study was to investigate the effect of ocean sound on symptoms in infants with infantile colic aged 0-3 months.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Diagnosis of infantile colic according to Wessel criteria
* The baby is born prematurely/maturely
* The baby is between 0-3 months
* Babies must have passed the newborn hearing screening test (the sound level used during the test is set at 30 decibels)
* Otoscopic examinations of babies should be performed by a specialist physician
* The baby has no diagnosis other than infantile colic on examination
* The baby does not have any chronic disease
* Mothers know how to read, write and speak Turkish
* No alternative application (massage, oil, herbal teas, etc.) should be used before the application

Exclusion Criteria:

* The baby has any acute and chronic disease
* The baby has a congenital anomaly
* The mother has diagnosed mental and psychological problems
* Diagnosis of lactose intolerance in infants by a physician
* Previously diagnosed with Infantile Colic and continuing medical treatment
* Babies have not passed the newborn hearing screening test
* Otoscopic examinations of infants not performed by a specialist physician

Ages: 0 Days to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
listening to ocean sounds reduces colic symptoms | babies in the intervention group will be played the sound of the ocean when crying for a week after the first encounter
  the sound of the ocean will be played to babies as an intervention. The effect of ocean sound on the infant's crying and sleep duration and infantile colic scale score will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: TÜLAY KUZLU AYYILDIZ, Study Director — ZONGULDAK BÜLENT ECEVİT ÜNİVERSİTESİ